CLINICAL TRIAL: NCT07181512
Title: Deep Learning-Based Opportunistic Screening of Coronary Artery Disease on Non-Contrast Chest CT: A Multicenter Study
Brief Title: Deep Learning CAD Screening on Chest CT
Acronym: CAD-AI
Status: Not yet recruiting | Type: Observational
Sponsor: Yifan Guo (Other Government)
Collaborators: Jinhua Municipal Central Hospital (Other); The Second Affiliated Hospital of Fujian Medical University (Other); First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor-Investigator, Yifan Guo, Lecturer, Department of Radiology, First Affiliated Hospital of Zhejiang Chinese Medical University, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Other Study IDs: CAD-AI-2025-V1.0
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis Stent
Keywords: Coronary Artery Disease; Non-contrast Chest CT; Coronary CT Angiography; Opportunistic Screening; Artificial Intelligence
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing non-contrast chest CT and CCTA: A cohort of patients who underwent both non-contrast chest CT and coronary CT angiography (CCTA) within 30 days. Clearly visualized coronary segments will be analyzed at the segment level for plaque composition and ≥50% stenosis using deep learning models. Both retrospective (2015-2024) and prospective (2025) cases are included.
  Interventions: Other: Deep Learning Analysis of Non-contrast Chest CT

INTERVENTIONS:
Other: Deep Learning Analysis of Non-contrast Chest CT — Analysis of clearly visualized coronary segments on non-contrast chest CT using deep learning models, compared with CCTA reference standard.

SUMMARY:
Coronary artery disease (CAD) is one of the leading causes of death worldwide. Many people have early atherosclerosis without symptoms, and some may develop significant coronary stenosis before any warning signs appear. Identifying high-risk individuals at an early stage is important to prevent heart attacks and other cardiovascular events.

Coronary CT angiography (CCTA) can directly evaluate plaque type and the degree of narrowing in the coronary arteries, but it is expensive, requires contrast injection, and involves higher radiation, making it unsuitable for large-scale screening. In contrast, non-contrast chest CT is widely used for health check-ups and lung disease follow-up. Such scans often provide clear views of certain coronary segments, which creates an opportunity to screen for CAD without additional cost or risk.

This multicenter study aims to develop and validate deep learning models to analyze coronary calcified segments that are visible on non-contrast chest CT. Two main objectives are: (1) to predict whether calcified segments contain mixed plaque components (both calcified and non-calcified); and (2) to predict whether these segments have significant narrowing (≥50% stenosis) as determined by CCTA. The study will also describe how often ≥50% stenosis is found in non-calcified segments, in order to demonstrate their low-risk nature.

The study includes retrospective data collected between 2015 and 2024, and a prospective external validation cohort starting in 2025. Approximately 1,417 patients with paired chest CT and CCTA have already been included for model development and testing. An additional 200 or more patients will be prospectively recruited for external validation.

This research may provide evidence that deep learning applied to routine non-contrast chest CT can serve as an opportunistic tool for early CAD risk screening in the general population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients who underwent both non-contrast chest CT and coronary CT angiography (CCTA) within 30 days
3. Coronary segments clearly visualized on non-contrast chest CT

Exclusion Criteria:

1. Segments with motion artifacts, metal artifacts, or stents preventing analysis
2. Vessel lumen completely obscured by calcification (unrecognizable vascular course)
3. Inability to match coronary segment location between non-contrast chest CT and CCTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non-contrast chest CT and CCTA, either during outpatient or inpatient clinical care, or as part of high-risk health examinations. Both retrospective cases (2015-2024) and prospectively recruited patients (2025) are included from five medical centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of plaque composition prediction | Baseline non-contrast chest CT to reference CCTA (within 30 days)
  Discrimination ability of the deep learning model to classify calcified coronary segments as purely calcified or mixed plaque, using CCTA as the reference standard. Evaluated with AUC, sensitivity, specificity.
Accuracy of ≥50% stenosis prediction | Baseline non-contrast chest CT to reference CCTA (within 30 days)
  Discrimination ability of the deep learning model to predict ≥50% luminal stenosis in calcified coronary segments, using CCTA as the reference standard. Evaluated with AUC, sensitivity, specificity, PPV, NPV.

SECONDARY OUTCOMES:
Incidence of ≥50% stenosis in non-calcified segments | Baseline non-contrast chest CT to CCTA (within 30 days)
  Descriptive statistics of ≥50% stenosis prevalence in non-calcified coronary artery segments.

IPD SHARING:
Plan to Share IPD: No
de-identified data available on reasonable request